CLINICAL TRIAL: NCT03558698
Title: Danish: Projekt God-Nat. Et Studie af søvnmiljøets Betydning for børns indlæringsevne English: Good Night: A Study of the Impact of the Sleep Environment on Learning in Children
Brief Title: Are Cognition and Sleep Affected by Exposure to Carbon Dioxide and Bio Effluents During Sleep?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 111017
Record Dates: First submitted 2018-05-16; First posted 2018-06-15 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-05

CONDITIONS: Cognitive Impairment, Mild; Sleep; Environmental Exposure
Keywords: cognition; sleep; carbon dioxide; bio effluents
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: The 36 children are divided into 6 groups of 6 children. Every group is exposed to all possible conditions (3) in a randomized order.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study is double-blinded but a few people in the research team are not blinded because of security reasons (they need to be able to control the concentrations of CO2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 (Other): * One night of good ventilation with a CO2 level of maximum 800 ppm
  * One night of good ventilation with high levels of CO2 (3000 ppm)
  * One night of poor ventilation with high concentrations of CO2 (3000 ppm) and other bio effluents (The order of the three conditions are randomized)
  Interventions: Other: Good ventilation; Other: Ventilation CO2; Other: Poor Ventilation
- Group 2 (Other): * One night of good ventilation with a CO2 level of maximum 800 ppm
  * One night of good ventilation with high levels of CO2 (3000 ppm)
  * One night of poor ventilation with high concentrations of CO2 (3000 ppm) and other bio effluents (The order of the three conditions are randomized)
  Interventions: Other: Good ventilation; Other: Ventilation CO2; Other: Poor Ventilation
- Group 3 (Other): * One night of good ventilation with High CO2 level of maximum 800 ppm
  * One night of good ventilation with high levels of CO2 (3000 ppm)
  * One night of poor ventilation with high concentrations of CO2 (3000 ppm) and other bio effluents (The order of the three conditions are randomized)
  Interventions: Other: Good ventilation; Other: Ventilation CO2; Other: Poor Ventilation
- Group 4 (Other): * One night of good ventilation with a CO2 level of maximum 800 ppm
  * One night of good ventilation with high levels of CO2 (3000 ppm)
  * One night of poor ventilation with high concentrations of CO2 (3000 ppm) and other bio effluents (The order of the three conditions are randomized)
  Interventions: Other: Good ventilation; Other: Ventilation CO2; Other: Poor Ventilation
- Group 5 (Other): * One night of good ventilation with a CO2 level of maximum 800 ppm
  * One night of good ventilation with high levels of CO2 (3000 ppm)
  * One night of poor ventilation with high concentrations of CO2 (3000 ppm) and other bio effluents (The order of the three conditions are randomized)
  Interventions: Other: Good ventilation; Other: Ventilation CO2; Other: Poor Ventilation
- Group 6 (Other): * One night of good ventilation with a CO2 level of maximum 800 ppm
  * One night of good ventilation with high levels of CO2 (3000 ppm)
  * One night of poor ventilation with high concentrations of CO2 (3000 ppm) and other bio effluents (The order of the three conditions are randomized)
  Interventions: Other: Good ventilation; Other: Ventilation CO2; Other: Poor Ventilation

INTERVENTIONS:
Other: Good ventilation — Good ventilation with a low concentration of CO2
Other: Ventilation CO2 — CO2 High and Good ventilation
Other: Poor Ventilation — Poor ventilation with high concentrations of CO2 and bio effluents

SUMMARY:
The aim of the project is to examine whether children's sleep and cognition are affected by exposure to CO2 and other bio effluents during sleep. The participants of the study are 36 children recruited from local schools in Aarhus, Denmark.

The study takes place in the climate chambers at the Department of Public Health, Aarhus University. These chambers allow for experimental testing on humans with advanced exposure generation while avoiding contamination from other sources and controlling temperature, humidity, noise, odor, and light.

The children will be sleeping in the chambers under three different conditions:

* One night of good ventilation with a CO2 level of maximum 800 ppm
* One night of good ventilation with high levels of CO2 (3,000 ppm)
* One night of poor ventilation with high concentrations of CO2 (3000 ppm) and other bio effluents.

The study is a within-group design, and groups of six children will be sleeping in the chambers for three nights (separated by seven days). The different groups of children are exposed to the conditions in a randomized order. The study is double-blinded (of security reasons the persons responsible for CO2 concentrations in the chambers are not blinded).

The study takes place on schools nights. The children arrive at 6 pm and leave for school the morning after. In the evening the children are tested for approximately 30-40 minutes to measure their cognitive performance using CANTAB (Cambridge Neuropsychological Test Automated Battery) on iPads. After completing the test, dinner is served and the children have some spare time before going to bed. During night, the quality of sleep (awake time and different sleep stages) will be monitored using Fitbit devices. Sleep quality will also be evaluated using a short sleep questionnaire. The next morning the cognitive performance of the children will be tested again using CANTAB before the children leave for school.

Our primary hypothesis is that children will perform worse on the cognitive test when exposed to high levels of CO2 and other bio effluents than compared to low levels of CO2 and bio effluents in a well-ventilated room. In addition to that our secondary hypotheses are:

* Children will perform worse on the cognitive test when exposed to high levels of CO2 and other bio effluents than compared to CO2 alone.
* Children will sleep less well in an environment with poor ventilation and high levels of CO2 and other bio effluents compared to sleeping in a well-ventilated room with low levels of CO2.
* Children will sleep less well in an environment with poor ventilation and high levels of CO2 and other bio effluents compared to sleeping in a room with high levels of CO2 alone.
* Children will sleep less well and perform worse on the cognitive test when exposed to high levels of CO2 compared to low levels of CO2.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children or children with a well-treated chronic disease not interfering with cognition and sleep quality
* Being able to accomplish a CANTAB test
* Completed questionnaires of sleep patterns

Exclusion Criteria:

* Unable to spend three nights (separated by seven days) in the climate chambers
* Conditions that prevent safe access to the chambers such as claustrophobia

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-06-22 (Actual)

PRIMARY OUTCOMES:
Reaction time (Simple) | 10 hours post start of exposure
  Reaction time in milliseconds. Outcome from CANTAB RTI Simple.

SECONDARY OUTCOMES:
CANTAB global composite score | 10 hours post start of exposure
  CANTAB global composite score = outcomes from CANTAB transformed into a global composite score.
Reaction Time (Five-Choice) | 10 hours post start of exposure
  Reaction time in milliseconds. Outcome from CANTAB RTI Five-Choice.
Sleep efficiency | Sleep measured for 9 hours during exposure in bed from 9 pm to 6 am.
  Sleep efficiency = Percentage of time in bed spent sleeping.

CONTACTS AND LOCATIONS:
Overall Officials: Torben Sigsgaard, Principal Investigator — Department of Public Health - Institute of Environmental and Occupational Medicine, Aarhus University
Locations (1):
- Aarhus University, Department of Public Health, Section for Environment, Occupation and Health, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No